CLINICAL TRIAL: NCT02886923
Title: Evaluation of Vision Effects of a Cosmetic Tinted Hydrogel Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-5856
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Results first posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Refractive Error
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Test/Control Sequence (Experimental): Subjects will wear the Hioxifilcon A Test contact lens and then the Hioxifilcon A with Cosmetic Ring Control contact lens for approximately three to four hours at each of the two measurement visits.
  Interventions: Device: Hioxifilcon A Test; Device: Hioxifilcon A With Cosmetic Ring Control
- Control/Test Sequence (Active Comparator): Subjects will wear the Hioxifilcon A with Cosmetic Ring Control contact lens and then the Hioxifilcon A Test contact lens for approximately three to four hours at each of the two measurement visits.
  Interventions: Device: Hioxifilcon A Test; Device: Hioxifilcon A With Cosmetic Ring Control

INTERVENTIONS:
Device: Hioxifilcon A Test — contact lens made with hioxifilcon A material
Device: Hioxifilcon A With Cosmetic Ring Control — contact lens made with hioxifilcon A material with a cosmetic ring on the lens

SUMMARY:
Subjects will wear 2 of 2 study contact lenses for a wearing time of approximately three to four hours at each of the visits in order to take measurements on binocular functional visual performance.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. The subject must be between 35 and 42 years of age (inclusive).
4. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -6.00 Diopters (D) to +4.00 D in each eye.
5. The subject's refractive cylinder must be ≤ 0.75 D in each eye.
6. The subject must have best corrected visual acuity of 20/30 or better in each eye.
7. The subject must be an adapted soft contact lens wearer in both eyes (defined as a minimum of 6 hours of Daily Wear (DW) for a minimum of 1 month prior to the study).
8. The subject must have normal eyes (i.e., no ocular medications or infections of any type).

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any ocular or systemic allergies or diseases that may interfere with contact lens wear.
3. Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV) by self-report.
4. Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
5. Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
6. Any ocular infection.
7. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, photorefractive keratectomy (PRK), laser-assisted in situ keratomileusis (LASIK), etc.)
8. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
9. Habitual contact lens type is toric, bifocal, in monovision contact lens wear, or is worn as extended wear.
10. Participation in any contact lens or lens care product clinical trial within 30 days prior to study enrollment.
11. Employee of investigational clinic (e.g., Investigator, Coordinator, Technician)

Ages: 35 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-01-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Optometry Technology Group, Ltd., London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 24 subjects were enrolled into this study. Of the enrolled subjects 23 were dispensed a study lens while 1 subject failed to meet all eligibility criteria. Of the dispensed subjects, all 23 completed the study.
Groups:
- Hioxilfilcon A (Test)/ Hioxifilcon A (Control): Subjects that received the Test lens during the first study period and the Control lens during the second study period.
- Hioxilfilcon A (Control)/ Hioxifilcon A (Test): Subjects that were received the Control lens during the first study period and the Test lens during the second stud period.
Period: Period 1
Arm/Group | Hioxilfilcon A (Test)/ Hioxifilcon A (Control) | Hioxilfilcon A (Control)/ Hioxifilcon A (Test)
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Hioxilfilcon A (Test)/ Hioxifilcon A (Control) | Hioxilfilcon A (Control)/ Hioxifilcon A (Test)
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dispensed Subjects: All subjects that were dispensed a study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.0 (2.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 14
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: Participants]
  United Kingdom | 23

OUTCOME MEASURES:

1. Primary Outcome: The Binocular Functional Visual Performance Under Distance Day Time Conditions (250 cd/m2) for Centrally Presented High Contrasts (HC) Time Controlled Visual Acuity (TCVA) Targets.
Description: Time Controlled Visual Acuity (TCVA) was assessed at 4 m using 250 cd/m2 luminance. The luminance requirements were same at the target and at the eye.
  Binocular functional visual performance was measured for the centrally presented high contrasts targets.
Time Frame: 15 minutes post lens fit
Population: All subjects who had successfully completed all required visits without any protocol deviations that the study responsible clinician documented as impacting the assessment of the hypotheses.
Measure: Mean (Standard Deviation); unit: -10 x logMAR
Groups:
- Hioxifilcon A (Test): Subjects that wore the Test lens in either the first or second period of the study.
- Hioxifilcon A (Control): Subjects that wore the Control lens in either the first or second period of the study.
Arm/Group | Hioxifilcon A (Test) | Hioxifilcon A (Control)
Number analyzed (Participants) | 23 | 23
-10 x logMAR | -0.03 (0.754) | 0.33 (0.656)

2. Secondary Outcome: The Binocular Functional Visual Performance Under Distance Night Time Conditions (2.5 cd/m2) for Centrally Presented HC TCVA Targets.
Description: Time Controlled Visual Acuity (TCVA) was assessed at 4 m using 2.5 cd/m2 luminance. The luminance requirements were same at the target and at the eye. Binocular functional visual performance was measured for the centrally presented high contrasts targets.
Time Frame: 15 Minutes post lens fitting
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: -10 x logMAR
Arm/Group | Hioxifilcon A (Test) | Hioxifilcon A (Control)
Number analyzed (Participants) | 23 | 23
-10 x logMAR | -2.16 (0.606) | -1.69 (0.727)

3. Secondary Outcome: The Binocular Functional Visual Performance Under Intermediate Vision Indoor Conditions (50 cd/m2) for Centrally Presented HC TCVA Targets.
Description: Time Controlled Visual Acuity (TCVA) was assessed at 67 cm using 50 cd/m2 luminance. The luminance requirements were same at the target and at the eye. Binocular functional visual performance was measured for the centrally presented high contrasts targets.
Time Frame: 15 Minutes post lens fitting
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: -10 x logMAR
Arm/Group | Hioxifilcon A (Test) | Hioxifilcon A (Control)
Number analyzed (Participants) | 23 | 23
-10 x logMAR | -1.29 (0.673) | -1.04 (0.782)

ADVERSE EVENTS:
Time Frame: Throughout the entire duration of the study. Approximately 8 weeks per subject.
Arm/Group | Hioxifilcon A (Test) | Hioxifilcon A (Control)
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-22): https://cdn.clinicaltrials.gov/large-docs/23/NCT02886923/Prot_SAP_000.pdf